CLINICAL TRIAL: NCT04586062
Title: Sponsor Initiated Expanded Access Protocol, Intermediate-Size Patient Population
Status: Available | Type: Expanded Access
Sponsor: Kedrion S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: SIEA-PLG
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Ligneous Conjunctivitis
MeSH Terms: conditions — Plasminogen Deficiency, Type I | interventions — Plasminogen

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Plasminogen — Human Plasminogen

SUMMARY:
The purpose of this protocol is to provide compassionate use of Kedrion Human Plasminogen Ophthalmologic Drops to an expanded population of patients diagnosed with ligneous conjunctivitis associated with type I Plasminogen deficiency until product licensure, and/or until a new clinical trial is available and the patients in treatment under Expanded Access are eligible to participate in the new trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with LC associated with Type I plasminogen deficiency, confirmed by laboratory documentation at screening visit, with or without ocular pseudomembranes. The presence of membranes in different areas is not an exclusion criterion.
* Subjects and their legally authorized representative, in the case of subjects <18 years of age, should be informed of the nature of the treatment, agree to its provision, sign and date the informed and data handling consent forms approved by the IRB.
* Subjects must be available for the duration of the treatment and agree to be compliant with the protocol visit and follow-up schedule.
* Subjects agree to keep the treating physician or specialist in charge informed about any occurrence related to the treatment.

Exclusion Criteria:

* Subjects with any condition which, in the opinion of the treating physician or specialist in charge might interfere with the treatment.
* Females of childbearing potential who are either pregnant or not using an adequate method of birth control (adequate is defined as hormonal contraceptive or partner vasectomy for at least 3 months, condoms, intrauterine device [IUD], abstinence or other prescribed birth control). Enrolled males must agree to utilize appropriate contraceptive methods to prevent pregnancy in partners.
* Females who are breastfeeding.

Sex: All
Age Groups: Child, Adult, Older Adult